CLINICAL TRIAL: NCT02008396
Title: A Placebo-controlled, Randomized, Blinded, Dose Finding Phase 2 Pilot Safety Study of MDMA-assisted Therapy for Social Anxiety in Autistic Adults
Brief Title: Phase 2 Pilot Safety Study of MDMA-assisted Therapy for Social Anxiety in Autistic Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lykos Therapeutics (Industry)
Collaborators: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MAA-1
Record Dates: First submitted 2013-12-06; First posted 2013-12-11 (Estimated); Results first posted 2020-10-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: Social Anxiety in Autistic Adults
Keywords: MDMA; autism; social anxiety
MeSH Terms: conditions — Autistic Disorder | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Inactive Placebo with Therapy (Placebo Comparator): Participants will receive inactive placebo during two psychotherapy sessions lasting approximately 7 hours.
  Interventions: Drug: Placebo; Behavioral: Therapy
- Group 1: MDMA-assisted therapy 75 mg/100mg (Experimental): Participants will receive 75 mg and 100 mg midomafetamine HCl during two sessions of MDMA-assisted therapy, respectively, lasting approximately 7 hours.
  Interventions: Drug: Midomafetamine HCl; Behavioral: Therapy
- Group 2: MDMA-assisted therapy 100 mg/125 mg (Experimental): Participants will receive 100 mg and 125 mg midomafetamine HCl during two sessions of MDMA-assisted therapy, respectively, lasting approximately 7 hours.
  Interventions: Drug: Midomafetamine HCl; Behavioral: Therapy

INTERVENTIONS:
Drug: Placebo — Subjects will receive capsules of lactose of identical appearance to MDMA capsules during each of two experimental sessions. Capsules will be administered along with therapy.
  Other Names: Inactive placebo
  Arms: Inactive Placebo with Therapy
Drug: Midomafetamine HCl — Participants in Group 1 receive 75 or 100 mg during the two experimental sessions and participants in Group 2 receive 100 or 125 mg during two experimental sessions.
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA
  Arms: Group 1: MDMA-assisted therapy 75 mg/100mg; Group 2: MDMA-assisted therapy 100 mg/125 mg
Behavioral: Therapy — Therapy conducted throughout experimental sessions. Therapists will use a largely nondirective approach. There will be periods of structured and unstructured interactions. The structured interactions will be selected based on elements of therapeutic interventions that are currently in use in this population for the treatment of social anxiety.
  Other Names: Manualized therapy

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is safe and effective at reducing social anxiety in adults with autism.

The main questions it aims to answer are:

* Do two sessions of MDMA-assisted therapy reduce social anxiety?
* What dose of MDMA is most effective at reducing social anxiety?

Researchers will compare two blinded sessions of MDMA-assisted therapy to two blinded sessions of placebo with therapy.

Participants will undergo three non-drug preparatory therapy sessions before the first blinded medication session. After each medication session, participants will undergo three non-drug integrative therapy sessions.

In Stage 2, participants who received placebo with therapy in the first two blinded sessions will be able to undergo two sessions with MDMA-assisted therapy.

DETAILED DESCRIPTION:
The main objective of this study was to collect safety data to examine whether MDMA-assisted therapy was tolerated and to estimate symptom reduction in social anxiety and other psychiatric symptoms that are common in the adult autistic population as evaluated by standard clinical measures. The primary outcome measure was change in social anxiety symptoms as measured by the Liebowitz Social Anxiety Scale (LSAS) [Heimberg et al., 1999].

Each of the 12 subjects participated in two blinded experimental sessions, with either MDMA or placebo, which lasted seven hours. Before experimental sessions, participants underwent three separate hour-long preparatory sessions to learn what to expect and complete pre-treatment assignments. After each experimental session, participants underwent three separate hour-long integrative sessions to help integrate their experiences and insights from the experimental sessions.

This study was designed as a dose escalation study to assist with the exploration of safety and finding the most effective dose in this population. Upon enrollment, participants (Group 1) were randomized to receive one dose of either placebo or 75 mg of midomafetamine HCl. In the second experimental session one month later, Group 1 subjects randomized to MDMA escalated to 100 mg of midomafetamine HCl, unless contraindicated. The second group of subjects enrolled (Group 2) were randomized to receive one dose of either placebo or 100 mg of midomafetamine HCl. In the second experimental session one month later, Group 2 subjects randomized to MDMA escalated to 125 mg of midomafetamine HCl, unless contraindicated.

The blind was maintained through the six-month follow-up. In Stage 2 after the blind was broken, subjects who received placebo in Stage 1 were offered an open-label extension with two experimental sessions of MDMA-assisted therapy scheduled one month apart. Subjects received 75 mg of midomafetamine HCl in the first session and escalated to 125 mg of midomafetamine HCl in the second session, unless contraindicated.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of Autism Spectrum Disorder.
* Have social anxiety.
* Are at least 21 years old.
* Have completed two years of college-level education or comparable vocational training.
* Are willing to refrain from psychiatric medication for at least 5 half-lives plus a week prior to experimental session.
* Agree to follow all study-related instructions and restrictions, including restrictions on food, alcohol and caffeine consumption prior to experimental sessions.
* Are willing to commit to preparatory sessions, medication management, experimental sessions, follow-up sessions and to complete evaluation instruments.
* Agree not to use MDMA/ecstasy outside of study sessions during the study, including the follow up period.
* Are willing to be contacted on a daily basis for a week after each experimental session.
* Are willing to provide a contact that is willing and able to be reached by investigators, accompany the subject during some or all of the study visits, and complete study measures.
* Are willing to give blood samples.
* Are proficient in speaking and reading English. Subjects communicating with text-to-speech technology will also be permitted to enroll.

Exclusion Criteria:

* Upon review of medical or psychiatric history must not have any current or past diagnosis that would be considered a risk to participation in the study.
* Are abusing illegal drugs.
* Are not able to give adequate informed consent.
* Are not able to attend face-to-face visits or those who plan to move out of the area within the treatment period.
* Are pregnant or nursing, or if are able to bear children and do not practice an effective means of birth control.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-04-11 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles S. Grob, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share outcome data appearing in any published reports upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Data and study-related documents will be available when all participants have completed the study
Access Criteria: Interested persons should correspond with the central contact for the study.

REFERENCES:
- [Background] Heimberg RG, Horner KJ, Juster HR, Safren SA, Brown EJ, Schneier FR, Liebowitz MR. Psychometric properties of the Liebowitz Social Anxiety Scale. Psychol Med. 1999 Jan;29(1):199-212. doi: 10.1017/s0033291798007879. PMID 10077308
- [Result] Danforth AL, Grob CS, Struble C, Feduccia AA, Walker N, Jerome L, Yazar-Klosinski B, Emerson A. Reduction in social anxiety after MDMA-assisted psychotherapy with autistic adults: a randomized, double-blind, placebo-controlled pilot study. Psychopharmacology (Berl). 2018 Nov;235(11):3137-3148. doi: 10.1007/s00213-018-5010-9. Epub 2018 Sep 8. PMID 30196397
- [Derived] Danforth AL, Struble CM, Yazar-Klosinski B, Grob CS. MDMA-assisted therapy: A new treatment model for social anxiety in autistic adults. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:237-49. doi: 10.1016/j.pnpbp.2015.03.011. Epub 2015 Mar 25. PMID 25818246
- See also: Link to open access copy of publication on study — http://link.springer.com/article/10.1007%2Fs00213-018-5010-9

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited by printed or internet advertisements, referrals from other health-care practitioners, and word-of-mouth. Potential participants were people, aged 21 or older, with a confirmed diagnosis of autism. The study was conducted at Los Angeles Biomedical Research Institute in Torrance, CA between February 2014 and October 2017.
Pre-assignment Details: One participant was excluded for not meeting eligibility criteria within exclusion window for enrollment.
Groups:
- Inactive Placebo With Psychotherapy: Subjects will receive inactive placebo during two psychotherapy sessions lasting approximately 7-8 hours.
- Group 1: MDMA-assisted Therapy 75mg/100mg: Participants will receive 75 mg midomafetamine HCl during their first MDMA-assisted therapy session and 100 mg midomafetamine HCl during their second MDMA-assisted therapy session.
- Group 2: MDMA-assisted Therapy 100mg/125mg: Participants will receive 100 mg midomafetamine HCl during their first MDMA-assisted therapy session and 125 mg midomafetamine HCl during their second MDMA-assisted therapy session.
Period: Stage 1
Arm/Group | Inactive Placebo With Psychotherapy | Group 1: MDMA-assisted Therapy 75mg/100mg | Group 2: MDMA-assisted Therapy 100mg/125mg
Started | 4 | 4 | 4
Completed (Primary Endpoint) | 3 | 4 | 4
Not Completed | 1 | 0 | 0
Period: Stage 2
Arm/Group | Inactive Placebo With Psychotherapy | Group 1: MDMA-assisted Therapy 75mg/100mg | Group 2: MDMA-assisted Therapy 100mg/125mg
Started | 3 | 0 | 0
Completed | 3 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set
Groups:
- Group 1 MDMA-assisted Therapy 75mg/100mg: Participants will receive 75 mg midomafetamine HCl during their first MDMA-assisted therapy session and 100 mg midomafetamine HCl during their second MDMA-assisted therapy session.
- Group 2 MDMA-assisted Therapy 100mg/125mg: Participants will receive 100 mg midomafetamine HCl during their first MDMA-assisted therapy session and 125 mg midomafetamine HCl during their second MDMA-assisted therapy session.
- Total: Total of all reporting groups
Arm/Group | Inactive Placebo With Psychotherapy | Group 1 MDMA-assisted Therapy 75mg/100mg | Group 2 MDMA-assisted Therapy 100mg/125mg | Total
Number analyzed (Participants) | 4 | 4 | 4 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.27 (3.77) | 37.93 (12.25) | 27.77 (5.87) | 31.32 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 2
  Male | 4 | 3 | 3 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 3 | 3
  Not Hispanic or Latino | 4 | 4 | 1 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Baseline Liebowitz Social Anxiety Scale (LSAS) Score [Mean (Standard Deviation); unit: units on a scale] | 83.3 (11.87) | 89.0 (8.60) | 94.5 (22.13) | 88.9 (14.67)

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS) Total Score 1-Month Post Experimental Session 2
Description: The LSAS is a 24-item, semi-structured interview on the severity of Social Anxiety Disorder. The LSAS separately assesses fear and avoidance of 24 social situations. The scale is divided into 2 subscales, 13 situations concerning performance anxiety, and 11 situations pertaining to social situations. The 24 items are first rated on a Likert Scale from 0 to 3 on fear felt during the situations, and then the same items are rated regarding avoidance of the situation. Combining the total scores for the Fear and Avoidance sections provides an overall score with a maximum of 144 points and a minimum of 0 points. The higher the score, the greater the anxiety symptoms. The overall scores are interpreted as: 55-65 is moderate, 65-80 is marked, 80-95 is severe, and greater than 95 is very severe social anxiety symptoms.
Time Frame: 1-Month Post Experimental Session 2
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Group 2: MDMA-assisted Therapy 100mg/125 mg: Participants will receive 100 mg midomafetamine HCl during their first MDMA-assisted therapy session and 125 mg midomafetamine HCl during their second MDMA-assisted therapy session.
Arm/Group | Group 1: MDMA-assisted Therapy 75mg/100mg | Group 2: MDMA-assisted Therapy 100mg/125 mg | Inactive Placebo With Psychotherapy
Number analyzed (Participants) | 4 | 4 | 3
score on a scale | 34.3 (10.41) | 55.5 (11.47) | 64.0 (13.34)

2. Primary Outcome: Change in Leibowitz Social Anxiety Scale (LSAS) Total Score From Baseline to 1-Month Post Experimental Session 2
Description: as for outcome 1
Time Frame: Baseline to 1-Month Post Experimental Session 2
Population: Safety Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Group 1: MDMA-assisted Therapy 75mg/100mg | Group 2: MDMA-assisted Therapy 100mg/125mg | Inactive Placebo With Psychotherapy
Number analyzed (Participants) | 4 | 4 | 3
score on a scale | -51.0 (8.19) | -39.0 (17.57) | -19.3 (18.77)

ADVERSE EVENTS:
Time Frame: All AEs from baseline to the end of stage 2 (approximately 10 months)
Description: Subjects counted once per event
Groups:
- Inactive Placebo With Psychotherapy (Stage 1): Subjects will receive inactive placebo during two psychotherapy sessions lasting approximately 7-8 hours.
Arm/Group | Group 1: MDMA-assisted Therapy 75mg/100mg | Group 2: MDMA-assisted Therapy 100mg/125mg | Inactive Placebo With Psychotherapy (Stage 1)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 1/4 | 4/4 | 1/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: MDMA-assisted Therapy 75mg/100mg (N=4) | Group 2: MDMA-assisted Therapy 100mg/125mg (N=4) | Inactive Placebo With Psychotherapy (Stage 1) (N=4)
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 1
Pain (General disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0
Ligament injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Retinal injury (Injury, poisoning and procedural complications) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
Depressed mood (Psychiatric disorders) | 0 | 2 | 0
Panic attack (Psychiatric disorders) | 0 | 1 | 0
Panic reaction (Psychiatric disorders) | 0 | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (3):
  • Study Protocol (2013-05-21): https://cdn.clinicaltrials.gov/large-docs/96/NCT02008396/Prot_002.pdf
  • Statistical Analysis Plan (2017-08-31): https://cdn.clinicaltrials.gov/large-docs/96/NCT02008396/SAP_001.pdf
  • Informed Consent Form (2015-07-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02008396/ICF_003.pdf